CLINICAL TRIAL: NCT05984069
Title: Impact of Frailty and ICU-AW on Post-ICU Fatigue Self-reported
Acronym: FICUF
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN962022/CHUSTE
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Post Intensive Care Syndrome
Keywords: Intensive Care Unit; frailty; fatigue; ICU acquired-weakness; FACIT-F; physical activity
MeSH Terms: conditions — postintensive care syndrome; Frailty; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients on etiologies: Patients over 18 admitted in ICU for all etiologies with mechanical ventilation over 5 days or length of stay in ICU over 10 days will be included
  Interventions: Other: observational prospective data collection

INTERVENTIONS:
Other: observational prospective data collection — Collection of data from medical records.

SUMMARY:
After a prolonged stay in Intensive Care Unit (ICU), fatigue is the most common symptom reported by patients in the Post Intensive Care Syndrome (PICS). Other complications have been described, including ICU-acquired weakness, leading to increased morbidity and mortality after discharge. Actually, risk factors associated with post-ICU fatigue self-reported are not really known.

DETAILED DESCRIPTION:
Frailty, defined as a decrease in physiological reserves leading to an alteration in the mechanisms of adaptation to stress, increases the incidence of PICS and could therefore be a cause of post-ICU fatigue self-reported.

The aim of this study is to identify a relationship between markers of frailty, ICU-AW, ICU story and the post-ICU fatigue self-reported 6 months discharge in patients with prolonged ICU stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a length of stay in intensive care > or equal to 7 days, or mechanical ventilation > or equal to 5 days

Exclusion Criteria:

* Scheduled surgery with admission in ICU
* Pregnancy
* Guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care, all etiologies combined, excluding immediate post-operative scheduled surgery, with mechanical ventilation for more than 5 days or length of stay in ICU over 10 days.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frailty | 1 year
  Relationship between frailty markers (CFS, IADL, sarcopenia and myosteatosis), ICU-AW, ICU story and post-ICU fatigue self-reported

SECONDARY OUTCOMES:
Fatigue | 1 year
  Prevalence of post-ICU fatigue self-reported 6 months discharge in prospective cohort
ICU-acquired weakness and fatigue | 1 year
  Correlation between post-ICU fatigue self-reported and muscular strength assessed by handgrip test
Fatigue, quality of life, anxiety and depressive disorder | 1 year
  Correlation between fatigue, quality of life, anxiety and depressive disorder
Kinetic of muscle mass loss and post-ICU fatigue self-reported | 1 year
  Correlation between the kinetic of muscle mass loss and post-ICU fatigue self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme MOREL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Chu Saint-Etienne, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No